CLINICAL TRIAL: NCT03964766
Title: Postoperative Pain Following Pulpectomy of Primary Molars With Rotary Instrumentation Versus Manual Instrumentation: A Randomized Clinical Trial
Brief Title: Pulpectomy of Primary Molars With Rotary Instrumentation Versus Manual Instrumentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Azhar Abdulrahman Ali Saleh Al-wesabi, phD student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200277
Record Dates: First submitted 2019-05-16; First posted 2019-05-28 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Chronic; Infection
Keywords: rotary files; Primary molar; Pulpectomy
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotary instrumentation (Experimental): endodontic treatment will be performed with the use of pedo rotary files that will be activated by engine
  Interventions: Device: Rotary instrumentation
- hand istrumentation (Active Comparator): endodontic treatment will be performed with the use of conventional hand files
  Interventions: Device: Hand instrumentation

INTERVENTIONS:
Device: Rotary instrumentation — using pedo rotary files in cleaning and shaping the root canals of infected primary molars
  Arms: rotary instrumentation
Device: Hand instrumentation — using conventional hand files in cleaning and shaping the root canals of infected primary molars
  Arms: hand istrumentation

SUMMARY:
One of the major concerns in pediatric dentistry is premature loss of necrotic primary teeth which may cause a deleterious effect on the growth of the facial skeletal complex. In order to sustain the primary tooth as a natural space maintainer, pulpectomy is considered the treatment of choice.

The essential part of endodontic treatment is to shape and clean the root canal effectively from infected tissue with microbial reduction, whilst maintaining the original configuration without creating any procedural errors . Even though, manual instrumentation as used for that purpose in deciduous teeth, presents some limitation concerning root canal cleaning, anatomical fidelity and chair-side time.

To achieve successful pulpectomy technique for the primary dentition in a fast and simple procedure, with short chair time as well as effective debridement of the root canals, rotary instrumentation is one of the methods recommended over the manual.

DETAILED DESCRIPTION:
1. Trial design:

   Randomized clinical trial, parallel groups design with 1:1 allocation ratio.
2. Method:

   Interventions

   A. Diagnostic procedure:
   * Clinical examination will be done on the dental clinic using mirror and probe to assess the eligibility.
   * Diagnosis of the cases will be performed according to guidelines of AAPD 2017 for treatment of vital pulp therapy in primary teeth.
   * An individual XCP (Extension Cone Paralleling) index will be prepared for each patient by registering the bite to allow consistent comparisons of the radiographs.
   * Preoperative periapical radiograph and photographs will be taken a baseline record.

   B. Intra operative procedure:
   * Local anesthesia administration using articaine 4% with epinephrine 1:100000.
   * Rubber dam application and access cavity preparation will be established using a sterile bur.
   * Coronal pulp tissue will be removed using sharp large spoon excavator.
   * Working length will be determined using no 15 hand K-file that will be kept 2mm short of radiographic apex.
   * Then, the root canal preparation will be done

     * In control group, hand instrumentation will be carried out using hand K-file up to no. 30 K-file using quarter turn and pull motion.
     * In intervention group, rotary instrumentation will be preceded by initial hand instrumentation using no. 15 K-file to check the patency. Then, the rotary instrumentation will be done using the Kedo-S rotary files for primary teeth with D1 and E1.
   * Using EDTA gel as a lubricating paste during canal preparation with rotary files.
   * Saline irrigation for removal of debris after each file.
   * Dryness will be done using paper points size 35 and 40.
   * Root canals will be obturated using calcium hydroxide iodoform paste (Metapex). The Metapex syringe willbe inserted into the root canal space, near the apex. The paste will be pressed down into the canals and the syringe will be slowly withdrawn.
   * The access cavity will be sealed using GC Fuji IX capsule.
   * The immediate postoperative radiograph will be done to reveal optimal filling with metapex.
   * After that, stainless steel crowns will be cemented by Ketac Cem.

   C. Follow up:

   Clinical and radiographic evaluation will be performed at 1week, 3, 6, 9 and 12 months.

   D. Criteria for discontinuing or modifying intervention:

   In case of unsuccessful outcomes of the intervention technique, the case will be managed .
3. Recruitment:

   Recruitment of the patients will be from the outpatient clinic of Pediatric Dentistry and Dental Public Health Department, Cairo University. Screening of patients will continue until the target population is achieved.
4. Implementation Co-supervisor; Fatma Korany will assign which participant tooth will be included to either control or intervention groups according to the generated random sequence.
5. Masking/blinding:

The radiographic outcomes assessor will be blinded in this study. 8- Data collection, management, and analysis: 9- Data collection methods

Baseline data will be collected by the operator through a paper-based Case Report custom made form (CRF) which will be developed by the research team. It will include the following items:

1. Patient serial number.
2. Demographic data.
3. Patients medical history:

   * Past medical history.
   * Any present disease or illness.
   * Current medication.
   * Any specific pre-treatment medication.
4. Past dental history.
5. Records for current dental condition (intra-oral examination and caries index). The custom made CRF will be developed before online registration of the study protocol. CRF will be anonymous where patients will be identified by their serial number. The full detailed personal data of the patient will be written in a separate sheet having the patient's serial number for further contact with patient, this sheet can be only seen by the operator and the supervisors. The Co-supervisor; Dr.Fatma Korany, will have the role to monitor the process of data collection and check if there is any incomplete CRF.

ELIGIBILITY:
Inclusion Criteria:

* Primary posterior teeth requiring pulpectomy.
* Cooperative patient in age range from 4 to 6 years
* Absence of internal or external pathologic root resorption.
* Presence of adequate coronal tooth structure.
* Two-thirds of each root remaining.
* Parent or guardian agree for participant in the study

Exclusion Criteria:

* Excessive mobility.
* Children lacking cooperative ability.
* Children with underlying systemic disease.
* Children with special health care needs.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain: modified wong-baker pain rating scale | 12 hours
  pain will be assessed using modified wong-baker pain rating scale (0-3),(zero)-no pain; ( one)-slight pain; (two)-moderate pain; and (three)-severe pain.
postoperative pain: modified wong-baker pain rating scale | 24 hours
  pain will be assessed using modified wong-baker pain rating scale (0-3),(zero)-no pain; ( one)-slight pain; (two)-moderate pain; and (three)-severe pain.
postoperative pain: modified wong-baker pain rating scale | 48 hours
  pain will be assessed using modified wong-baker pain rating scale (0-3),(zero)-no pain; ( one)-slight pain; (two)-moderate pain; and (three)-severe pain.
Postoperative pain: modified wong-baker pain rating scale | 72 hours
  pain will be assessed using modified wong-baker pain rating scale (0-3),(zero)-no pain; ( one)-slight pain; (two)-moderate pain; and (three)-severe pain.

SECONDARY OUTCOMES:
Tenderness to percussion | Up to 1 year
  Percussion test ,Binary (+/-)
Fistula | Up to 1 year
  Visual examination by operator,Binary (+/-)
Instrumentation time | 15 Minutes
  The time spent using both techniques will be measured and compared between the groups. The time will be recorded in minutes using a stopwatch since the beginning of instrumentation until the beginning of restorative procedure.
Furcation or periapical radiolucency | 6 month
  Digital Radiograph ,Binary (+/-)
Furcation or periapical radiolucency | 12 month
  Digital Radiograph ,Binary (+/-)

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Abdelgawad, PhD, Study Director — Lecturer of Pediatric Dentistry; Kamal El Motayam, PhD, Study Chair — Professor of Pediatric Dentistry

IPD SHARING:
Plan to Share IPD: Yes
after thesis defense. the study will be published internationally to be available for everyone
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: study will be available within 2 year.
Access Criteria: Not yet

REFERENCES:
- [Background] Panchal V, Jeevanandan G, Subramanian E. Comparison of instrumentation time and obturation quality between hand K-file, H-files, and rotary Kedo-S in root canal treatment of primary teeth: A randomized controlled trial. J Indian Soc Pedod Prev Dent. 2019 Jan-Mar;37(1):75-79. doi: 10.4103/JISPPD.JISPPD_72_18. PMID 30804311
- [Background] Makarem A, Ravandeh N, Ebrahimi M. Radiographic assessment and chair time of rotary instruments in the pulpectomy of primary second molar teeth: a randomized controlled clinical trial. J Dent Res Dent Clin Dent Prospects. 2014 Spring;8(2):84-9. doi: 10.5681/joddd.2014.015. Epub 2014 Jun 11. PMID 25093051
- [Background] Panchal V, Jeevanandan G, Subramanian EMG. Comparison of post-operative pain after root canal instrumentation with hand K-files, H-files and rotary Kedo-S files in primary teeth: a randomised clinical trial. Eur Arch Paediatr Dent. 2019 Oct;20(5):467-472. doi: 10.1007/s40368-019-00429-5. Epub 2019 Mar 12. PMID 30864090
- See also: Pinheiro, S., Santos, N. & Imparato, J. (2012) Analysis of the instrumentation time and cleaning between manual and rotary techniques in deciduous molars. Rsbo, 9 (3), pp.238-244. — https://pdfs.semanticscholar.org/cce0/6b2e5908ce798bdef7dce74421d5f5e7257f.pdf
- See also: Ochoa-Romero, T., Veronica Mendez-Gonzalez, H.F.-R. & Pozos-Guillen, A.J. (2011) Comparison Between Rotary and Manual Techniques on Duration of Instrumentation and Obturation Times in Primary Teeth. — https://www.ncbi.nlm.nih.gov/pubmed/22046692